CLINICAL TRIAL: NCT06623474
Title: Correlation Study of Lipid Metabolites as Markers of Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2024-361
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients diagnosed with hepatocellular carcinoma: Patients diagnosed with hepatocellular carcinoma according to the guidelines for the diagnosis of primary liver cancer
  Interventions: Diagnostic Test: diagnosed by traditional diagnostic markers（such as AFP or CT etc.）
- Patients diagnosed with non-hepatocellular carcinoma otherwise requiring hepatic resection: Patients who can be excluded from the diagnosis of hepatocellular carcinoma according to the guidelines for the diagnosis of primary liver cancer but required hepatic resection for other liver diseases
  Interventions: Diagnostic Test: diagnosed by traditional diagnostic markers（such as AFP or CT etc.）

INTERVENTIONS:
Diagnostic Test: diagnosed by traditional diagnostic markers（such as AFP or CT etc.） — A prospective observational cohort study to explore the advantages of lipid metabolites as diagnostic markers for hepatocellular carcinoma compared to traditional diagnostic markers for hepatocellular carcinoma (e.g., AFP, enhanced CT, etc.).
  Other Names: diagnosed by lipid metabolites

SUMMARY:
As one of the common malignant tumors in China, primary liver cancer, whose incidence rate and mortality rate are always in the top five, is seriously threatening the health of people. Therefore, early diagnosis and treatment of primary liver cancer are of great significance. In recent years, the incidence of primary liver cancer, which is caused by hepatic steatosis or metabolic dysfunction-related liver disease, is increasing year by year, and it has become one of the fastest rising causes in some developed countries. More and more studies have also confirmed that the levels of different kinds of lipids and their metabolites are correlated with the development of hepatocellular carcinoma. In this study, the researchers performed qualitative and quantitative analyses of various common lipid metabolites in plasma and liver cancer tissues of hepatic resection patients with hepatocellular carcinoma, collected tumor-related pathological data from the patients, and investigated the correlation between the lipid metabolites and the development of hepatocellular carcinoma, in order to provide a new idea for the early diagnosis and treatment of primary hepatocellular carcinoma, as well as for screening of hepatocellular carcinoma markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years old undergoing hepatic resection for hepatocellular carcinoma (diagnostic criteria for hepatocellular carcinoma refer to the guidelines for the diagnosis and treatment of primary hepatocellular carcinoma).
* Voluntary signing of informed consent

Exclusion Criteria:

* In the judgment of the investigator, they are not suitable to participate in this study.
* Patients with hepatic malignant tumors with invasion of the main portal vein and its first-order branches, the common hepatic duct and its first-order branches, the main hepatic vein and the inferior vena cava, or extrahepatic metastases.
* Surgery with biliary tract exploration or reconstruction in the presence of biliary obstruction.
* Surgery combined with splenectomy or splenic artery ligation
* Preoperative combination of cardiac, pulmonary, renal and other organs with major underlying diseases.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-80 years old undergoing hepatic resection for hepatocellular carcinoma (diagnostic criteria for hepatocellular carcinoma refer to the guidelines for the diagnosis and treatment of primary hepatocellular carcinoma).
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2032-06-30 (Estimated); Study Completion 2032-07-01 (Estimated)

PRIMARY OUTCOMES:
Lipid Metabolite Levels | Pre-operative and 1, 3 and 5 days post-operatively
  Lipids are extracted in the laboratory and sent to specialized laboratories for LC/MS non-targeted lipidomic assays to measure lipid metabolite levels in plasma and tissues.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lei Y, Xie C, Mo X, Zhuang B, Li Q, Liu C, Liao L, Wang B, Zeng M, Tang S, Liu H, Xiao Y, Li S, Cai D, Li C, Zhou J, Li J, Li Y, Wang K. Preoperative plasma ceramide profiling coupled with machine learning accurately predicts recurrence of hepatocellular carcinoma after resection. Lipids Health Dis. 2025 Nov 6;24(1):355. doi: 10.1186/s12944-025-02749-6. PMID 41194075